CLINICAL TRIAL: NCT06591741
Title: Effects of Dietary Protocatechuic Acid (PCA) on the Function and Structure of Participants With Knee Prosthetic Joint Infection (PJI) as Measured by Standard Biomarkers
Brief Title: PCA Administration in Prosthetic Joint Infection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Dean Reeves Clinic (Other)
Collaborators: Lanny Johnson, M.D. (Unknown); Leo Whiteside, M.D. (Unknown)
Responsible Party: Principal Investigator, Dr. Dean Reeves, Primary Investigator, Dr. Dean Reeves Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PCAinPJI-01
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Prosthetic Joint Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PCA administraton (Other)
  Interventions: Dietary Supplement: Oral PCA

INTERVENTIONS:
Dietary Supplement: Oral PCA — PCA 1,000 mg BID until surgery, held until anticoagulation, and resumed at 1,000 mg daily for 4 years

SUMMARY:
Determine if dietary protocatechuic acid (PCA) will affect health biomarkers in patient undergoing revision surgery for a knee prosthetic joint infection

DETAILED DESCRIPTION:
Patients who are scheduled to undergo revision surgery for a knee prosthetic joint infection are given PCA prior to surgery for a time period determined by a previous pilot study. PCA is then post-operatively until anticoagulation is stopped, and then will be resumed for four years post revision surgery. Measurement of changes in glucose control, immunity, will be measured over the first 3 months post-revision, and the post-revision reinfection rate over the full 4 years will be compared to a cohort rate

ELIGIBILITY:
Inclusion Criteria:

* 3 weeks or more after total knee arthroplasty
* One or more symptoms of infection, including redness, swelling, pain, increasing range of motion loss, fever, nausea, and loss of appetite.
* WBC count of aspirate >50,000 cells per μL

Exclusion Criteria:

* Not willing to undergo blood draw at 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in immunity factor CXCL9 from 0 to 3 months | 0 and 3 months
Change in HbA1c from 0 to 3 months | 0 and 3 months

SECONDARY OUTCOMES:
Reinfection rate after revision for prosthetic joint infection | 0 to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D Reeves, M.D., Principal Investigator — K. Dean Reeves, M.D., P.A.